CLINICAL TRIAL: NCT03181763
Title: Evaluation of 3,4-methylenedioxymethamphetamine (MDMA) on Startle Response
Brief Title: Evaluation of MDMA on Startle Response
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MPVA-4
Record Dates: First submitted 2017-06-05; First posted 2017-06-09 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Startle Response
Keywords: MDMA; Startle response; sleep; Oxytocin
MeSH Terms: interventions — Lactose; N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Intervention Model Description: Blinded, placebo between group; all participants undergo fear conditioning, with half randomized to receive 100 mg MDMA and half receiving inactive placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 100 mg MDMA HCl (Experimental): Participants receive 100 mg MDMA HCl on their second visit
  Interventions: Drug: Midomafetamine; Behavioral: Acoustic startle
- Placebo (Placebo Comparator): Participants receive inactive placebo on their second visit
  Interventions: Drug: Placebo; Behavioral: Acoustic startle

INTERVENTIONS:
Drug: Placebo — Participants will receive inactive placebo on their second visit.
  Other Names: inactive placebo; lactose
  Arms: Placebo
Drug: Midomafetamine — Participants will receive 100 mg midomafetamine HCl on their second visit
  Other Names: 3,4-methylenedioxymethamphetamine; MDMA; midomafetamine HCl
  Arms: 100 mg MDMA HCl
Behavioral: Acoustic startle — Startle assessment
  Other Names: startle test

SUMMARY:
The goal of this clinical trial is to learn if MDMA impacts startle response in healthy participants.

The main question it aims to answer is: Does MDMA impact participant's performance on a startle test?

Researchers will compare healthy volunteers who have taken MDMA to those who have taken placebo.

Participants will first undergo a 1-hour startle test. The next day, they will be randomized to receive either MDMA or placebo followed by another startle test and vitals signs and blood measurements. Participants will return the next day for a final startle test. Their sleep will be tracked by a Fitbit device.

DETAILED DESCRIPTION:
This is a randomized, blinded, placebo-controlled Phase 1 study that aims to evaluate the impact of 3,4-methylenedioxymethamphetamine (MDMA) on startle response.

This study will enroll healthy participants. At Visit 1, all participants will undergo a 1-hour startle test. Acoustic startle will be measured through assessing eye-blink response from the orbicularis oculi muscles in response to a 106 dB noise, using sensors under the eye. While watching the computer monitor, the participant will also experience several brief blasts of air directed at the throat.

At Visit 2 (24 hours later), participants will be randomized to receive 100 mg of MDMA or inactive placebo, after which they will undergo another startle test. Participants enrolled in the study who agree to do this will have their blood drawn to measure levels of oxytocin, and possibly other hormones or proteins, such as cortisol or brain-derived neurotrophic factor (BDNF). Measuring oxytocin will be blind to condition, and the decision will happen before randomization to either condition. Blood will be drawn before MDMA or placebo administration, and eight times afterwards.The researchers will measure pulse, blood pressure and temperature once before and six times after receiving MDMA or placebo, and study participants will complete a questionnaire about their experience.

At Visit 3, participants will return for a final startle test and recall task. Sleep will be measured via self-report and Fitbit during study participation.

ELIGIBILITY:
Inclusion Criteria:

* Persons aged 21 to 55.
* Ability to visually read and understand English language.
* Live within in metro Atlanta area
* Previously used MDMA in a recreational or research setting
* If a person is of childbearing potential (able to bear children), they must have a negative pregnancy test at study entry and prior to the Experimental Session. They must agree to use adequate birth control through 10 days after the last dose of MDMA. Adequate birth control methods include intrauterine device (IUD), injected or implanted hormonal methods, abstinence, oral hormones plus a barrier contraception or double barrier contraception. Two forms of contraception are required with any barrier method or oral hormones (i.e. condom plus diaphragm, condom or diaphragm plus spermicide, oral hormonal contraceptives plus spermicide or condom). Not of childbearing potential is defined as permanent sterilization, postmenopausal, or male.
* (For sub-study measuring serum oxytocin) Willing to have periodic blood draws

Exclusion Criteria:

* Upon review of medical or psychiatric history, have any current or past diagnosis that would be considered a risk to participating in the study.
* Are abusing illegal drugs.
* Current use of any psychoactive medications, including antidepressants, mood stabilizers, sedatives, stimulants, antipsychotics, anxiolytics, or beta-blockers
* Are not able to give adequate informed consent.
* Uncontrolled hypertension, or clinically significant cardiac arrhythmia, as detected by electrocardiogram.
* Currently pregnant or breast-feeding.
* History of acute angle glaucoma.
* Hearing impairment as assessed by audiometer; unable to detect tones below 40 dB in right or left ear.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
EMG of right orbicularis oculi muscle | Four days post-enrollment
  Description: Measure of startle response to noise after fear extinction training

SECONDARY OUTCOMES:
Systolic blood pressure pre-drug | 5 minutes pre-drug
  Systolic blood pressure measured prior to administration of MDMA or placebo
Systolic blood pressure 45 min post-drug | 45 minutes post-drug
  Systolic blood pressure measured 45 minutes after MDMA or placebo administration
Systolic blood pressure 1 h 15 min post-drug | 1 hour 15 minutes post drug
  Systolic blood pressure measured 1 hour 15 minutes after MDMA or placebo administration
Systolic blood pressure 1 h 45 min post-drug | 1 hour 45 minutes post drug
  Systolic blood pressure measured 1 hour 45 minutes after MDMA or placebo administration
Systolic blood pressure 3 h post-drug | 3 hours post-drug
  Systolic blood pressure measured 3 hours after MDMA or placebo administration
Systolic blood pressure 4 h post-drug | 4 hours post-drug
  Systolic blood pressure measured 4 hours after MDMA or placebo administration
Systolic blood pressure 5 h post-drug | 5 hours post-drug
  Systolic blood pressure measured 5 hours after MDMA or placebo administration
Systolic blood pressure 6 h post-drug | 6 hours post-drug
  Systolic blood pressure measured 6 hours after MDMA or placebo administration
Diastolic blood pressure pre-drug | 5 minutes pre-drug
  Diastolic blood pressure measured prior to MDMA or placebo administration
Diastolic blood pressure 45 min post-drug | 45 minutes post-drug
  Diastolic blood pressure measured 45 minutes after MDMA or placebo administration
Diastolic blood pressure 1 h 15 min post-drug | 1 hour 15 minutes post-drug
  Diastolic blood pressure measured 1 h 15 minutes after MDMA or placebo administration
Diastolic blood pressure 1 h 45 min post-drug | 1 hour 45 minutes post drug
  Diastolic blood pressure measured 1 h 45 minutes after MDMA or placebo administration
Diastolic blood pressure 3 h post-drug | 3 hours post-drug
  Diastolic blood pressure measured 3 hours after MDMA or placebo administration
Diastolic blood pressure 4 hours post-drug | 4 hours post-drug
  Diastolic blood pressure measured 4 hours after MDMA or placebo administration
Diastolic blood pressure 5 hours post-drug | 5 hours post-drug
  Diastolic blood pressure measured 5 hours after MDMA or placebo administration
Diastolic blood pressure 6 hours post-drug | 6 hours post-drug
  Diastolic blood pressure measured 6 hours after MDMA or placebo administration
Pulse pre-drug | 5 minutes pre-drug
  Pulse (assessing heart rate) measured prior to MDMA or placebo administration
Pulse 45 min post-drug | 45 minutes post-drug
  Pulse (assessing heart rate) measured 45 min after MDMA or placebo administration
Pulse 1 h 15 min post-drug | 1 hour 15 minutes post-drug
  Pulse (assessing heart rate) measured 1 hour 15 min after MDMA or placebo administration
Pulse 1 h 45 min post-drug | 1 hour 45 minutes post-drug
  Pulse (assessing heart rate) measured 1 hour 45 min after MDMA or placebo administration
Pulse 3 h post-drug | 3 hours post-drug
  Pulse (assessing heart rate) measured 3 hours after MDMA or placebo administration
Pulse 4 h post-drug | 4 hours post-drug
  Pulse (assessing heart rate) measured 4 hours after MDMA or placebo administration
Pulse 5 h post-drug | 5 hours post-drug
  Pulse (assessing heart rate) measured 5 hours after MDMA or placebo administration
Pulse 6 h post-drug | 6 hours post-drug
  Pulse (assessing heart rate) measured 6 hours after MDMA or placebo administration
Body temperature pre-drug | 5 minutes pre-drug
  Body temperature measured before MDMA or placebo administration
Body temperature 45 minutes post-drug | 45 minutes post-drug
  Body temperature measured 45 minutes after MDMA or placebo administration
Body temperature 1 h 15 minutes post-drug | 1 hour 15 minutes post-drug
  Body temperature measured 1 hour 15 minutes after MDMA or placebo administration
Body temperature 1 h 45 minutes post-drug | 1 hour 45 minutes post-drug
  Body temperature measured 1 hour 45 minutes after MDMA or placebo administration
Body temperature 3 hours post-drug | 3 hours post-drug
  Body temperature measured 3 hours after MDMA or placebo administration
Body temperature 4 hours post-drug | 4 hours post-drug
  Body temperature measured 4 hours after MDMA or placebo administration
Body temperature 5 hours post-drug | 5 hours post-drug
  Body temperature measured 5 hours after MDMA or placebo administration
Body temperature 6 hours post-drug | 6 hours post-drug
  Body temperature measured 6 hours after MDMA or placebo administration
Plasma oxytocin (OT) levels predrug | 5 min prior to drug administration
  In people who agree to it, blood collected to assess levels of oxytocin prior to MDMA or placebo administration on day of drug administration
Plasma oxytocin (OT) levels 5 min post-drug | 5 min post-drug administration
  In people who agree to it, blood collected to assess levels of oxytocin approximately 5 minutes after MDMA or placebo administration
Plasma oxytocin (OT) levels 20 min post-drug | 20 min post-drug administration
  In people who agree to it, blood collected to assess levels of oxytocin approximately 20 minutes after MDMA or placebo administration
Plasma oxytocin (OT) levels 95 min post-drug | 95 min post-drug administration
  In people who agree to it, blood collected to assess levels of oxytocin approximately 95 minutes (approximately 1.5 h) after MDMA or placebo administration
Plasma oxytocin (OT) levels 110 min post-drug | 110 min post-drug administration
  In people who agree to it, blood collected to assess levels of oxytocin approximately 110 minutes after MDMA or placebo administration
Plasma oxytocin (OT) levels 185 min post-drug | 185 min post-drug administration
  In people who agree to it, blood collected to assess levels of oxytocin approximately 185 minutes after MDMA or placebo administration
Plasma oxytocin (OT) levels 200 min post-drug | 200 min post-drug administration
  In people who agree to it, blood collected to assess levels of oxytocin approximately 200 minutes after MDMA or placebo administration
Plasma oxytocin (OT) levels 240 min post-drug | 240 min post-drug administration
  In people who agree to it, blood collected to assess levels of oxytocin approximately 240 minutes after MDMA or placebo administration
Plasma oxytocin (OT) levels 300 min post-drug | 300 min post-drug administration
  In people who agree to it, blood collected to assess levels of oxytocin approximately 300 minutes after MDMA or placebo administration

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Rothbaum, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maples-Keller JL, Norrholm SD, Burton M, Reiff C, Coghlan C, Jovanovic T, Yasinski C, Jarboe K, Rakofsky J, Rauch S, Dunlop BW, Rothbaum BO. A randomized controlled trial of 3,4-methylenedioxymethamphetamine (MDMA) and fear extinction retention in healthy adults. J Psychopharmacol. 2022 Mar;36(3):368-377. doi: 10.1177/02698811211069124. Epub 2022 Feb 15. PMID 35166140